CLINICAL TRIAL: NCT06785285
Title: Comparative Study of Fentanyl vs Dexmedetomidine as Adjuvants to Intrathecal Bupivacaine in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nehal Samir Esmail, Lecturer of Anesthesia, intensive care and pain management Faculty of Medicine, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Nehal Samir
Record Dates: First submitted 2024-11-27; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-03

CONDITIONS: Cesarean Section
MeSH Terms: interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): About 30 patients received Dexmeditomidine 5 ug and added to it 10 mg hyperbaric bupivicaine 0.5 % .
  Interventions: Drug: Dexmedetomidine
- Group B (Active Comparator): About 30 patients received fentanyl 25 ug and added to it 10 mg hyperbaric bupivicaine 0.5 % .
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — To compare the effects of fentanyl and dexmedetomidine when used as adjuvants to intrathecal bupivacaine in elective cesarean section, assessing their impact on the onset and duration of spinal anesthesia, quality of analgesia, hemodynamic stability, incidence of side effects, and neonatal outcomes
  Other Names: fentanyl 25 ug

SUMMARY:
The quality of the spinal anesthesia has beenreported to be improved by the addition of opioids (such as morphine, fentanyl and sufentanil) and other drugs (such as dexmedetomidine, clonidine, magnesium sulfate (Mg), neostigmine, ketamine, and midazolam).

Opioids such as fentanyl in combination with bupivacaine improvesthe quality of intraoperative and early postoperative subarachnoid block. Although, fentanylensures superior quality of analgesia, it is associated with many side effects. This has directed theresearch toward the use of newer and betteradjuvants for spinal anesthesia such as clonidineand dexmedetomidine

DETAILED DESCRIPTION:
Spinal anesthesia is still the first choice for cesarean section due to its deep sensoryblock as well as fewer side effects on mother and fetus. Despite many benefits ofthismethod, it has a short duration and cannot provide sufficient postoperativeanalgesia.Adequate postoperative analgesia plays a crucial role in cesarean delivery because itallows better breastfeeding and caring for newborns.

Dexmedetomidine is a relatively newer highly selectivealpha-2 adrenoceptor agonist agent that producesanalgesic and sedative effects. It has also been used asan adjuvant in Spinal anesthesia resulting in prolonged duration ofblock and improved postoperative analgesia without anyassociated hypotension or other adverse events

Fentanyl is a synthetic opioid with central action,which is used widely for pain control. Intrathecal fentanyl is usually added to other local anesthetics to increase anesthesia and analgesia. It has improved spinal anesthesia and reduced the anesthetic drug-related side effects including pruritus,nausea, and vomiting.

Adjuvant drugs added to the intrathecal bupivacaine can decrease the dose of local anesthetics and guarantee sensory and motor block. Intrathecal adjuvants include fentanyl and dexmedetomidine as receptor agonists, which have sedative, analgesic, perioperative sympatholytic, anesthetic-sparing, and hemodynamic-stabilizing properties.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the childbearing period
* aged 18 to 40 years
* Gestational age ≥37 weeks of pregnancy
* ASA I and II candidates for elective cesarean section under spinal anesthesia.

Exclusion Criteria:

* The patients with emergency conditions,
* Contraindication of spinal anesthesia,
* History of valvular heart disease,
* History of allergy or sensitivity to applied drugs and
* Patients with placenta previa
* Failed blockade or need for induction of general anesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Pain Relief | from 0 hours to 6 hours after the procedure
  Patient's pain score will be assessed using visual analogue scale (VAS); scored from 0-10 (where 0=no pain and 10=the worst pain imaginable) during the recovery room (T0) and at one, three, and six hours (T1, T3, and T6) in the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Nehal samir esmail, Lecturer, Principal Investigator — Sohag University, Faculty of medicine
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No